CLINICAL TRIAL: NCT00392028
Title: Penetration of Ertapenem Into Bone in Patients With Diabetes Mellitus or Peripheral Vascular Diseases Who Underwent Bellow Knee Amputation
Brief Title: Penetration of Ertapenem Into Bone
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no recruitment
Sponsor: HaEmek Medical Center, Israel (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: p1101v1
Record Dates: First submitted 2006-10-24; First posted 2006-10-25 (Estimated); Last update posted 2007-07-13 (Estimated); Status verified 2007-07

CONDITIONS: Amputation
Keywords: Ertapenem; Bone drug level; Blood drug level; Tissue drug level
MeSH Terms: interventions — Ertapenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ertapenem

SUMMARY:
The aim of the study is to determine the penetration levels of ertapenem into bone tissues in patients with Diabetes Mellitus (D.M) or Peripheral Vascular Diseases (P.V.D) undergoing amputation, and to correlate theme to the concentration of the drug in blood and other soft tissues

DETAILED DESCRIPTION:
Twelve patients with D.M or P.V.D who are undergoing bellow knee amputation with or without gangrene.

Within four weeks prior the amputation a vascular profile will be determined by Doppler and skin perfusion will be determined by transcutaneous oxygen pressure measurements (TcPO2) on the dorsal side of the mid foot of the affected limb.

Each patient will receive 1 g of Ertapenem in 100 ml of normal saline by IV infusion -during 30 minutes through IVAC:

* -2 days prior the amputation
* -1 day prior the amputation
* 1 hour before amputation The infusions will be started approximately at the same time of the 3rd infusion, prior the planned amputation.

Blood samples (approximately 6ml each) will be collected before Ertapenem administration, simultaneously with bone and soft tissue samples at the time of amputation and at the end of the surgery

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Diabetes Mellitus or Peripheral Vascular Disease
* Undergoing bellow knee amputation with or without gangrene
* Patients without clinical signs of acute infection
* Creatinine Clearence more than 60 cc/ min

Exclusion Criteria:

* Known hypersensitivity to any component of ertapenem or to other drugs in the same class.
* Patients who have demonstrated anaphylactic reactions to beta-lactams.
* CNS disorders (e.g., brain lesions or history of seizures).
* Patient treated with other antibiotics at least 72 hours.
* Pregnant women, nursing women, or fertile women not practicing adequate methods of contraception.
* Patient or legal representative of the patient is unable to provide written informed consent for any reason.
* Patient has a history of any illness that, in the opinion of the investigator, might confound the results of the study or pose additional risk in administering the study drug to the patient.
* Neutropenia
* Renal failure
* Hepatic Insufficiency: > x 2 upper limit.
* A need for any additional concomitant systemic antibacterial agent.
* Life expectancy less than 6 month
* Patient is undergoing immunosuppressive therapy, including use of high dose corticosteroids (e.g.,20 mg or more prednisone or equivalent per day)
* Patient is in a situation or has a condition which, in the investigator's opinion, may interfere with optimal participation in the study.
* Participation in an another clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2006-11; Study Completion 2007-07 (Estimated)

PRIMARY OUTCOMES:
blood,tissue and bone drug levels | 3 days each patient

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Kitzes, Study Director — Clinical Pharmacology Unit, Carmel Medical Center, Haifa
Locations (2):
- Israel (2):
  - Ha'Emek Medical Center, Afula
  - Haemek Medical Center INFECTIOUS DISEASES UNIT, Afula